CLINICAL TRIAL: NCT05413382
Title: A Randomized, Double-Blind, Crossover, Clinical Study to Investigate the Effect of an Investigational Lozenge (Biofresh® 4plus) Versus Placebo Control on Oral Malodor (Intra-Oral Halitosis)
Brief Title: Effect of an Investigational Lozenge (Biofresh® 4plus) Versus Placebo Control on Oral Malodor (Intra-Oral Halitosis)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novozymes A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: NZ-OHBF-2021-02
Record Dates: First submitted 2021-10-05; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2021-10

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational lozenge (Active Comparator): Lozenge containing the enzyme polyphenol oxidase and green coffee extract
  Interventions: Dietary Supplement: Biofresh® 4plus
- Placebo lozenge (Placebo Comparator): Lozenge equal to active comparator but without active ingredients
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Biofresh® 4plus — Participants will be instructed to use their assigned lozenge three times per day for seven days, preferably after breakfast, lunch, and dinner meals and to avoid eating and drinking for 30 minutes after consuming the lozenge.
  Arms: Investigational lozenge
Dietary Supplement: Placebo — Participants will be instructed to use their assigned lozenge three times per day for seven days, preferably after breakfast, lunch, and dinner meals and to avoid eating and drinking for 30 minutes after consuming the lozenge.
  Arms: Placebo lozenge

SUMMARY:
This study is designed to evaluate the effect of an investigational lozenge with the enzyme polyphenol oxidase and green coffee extract in reducing and controlling intra-oral halitosis following immediate use and daily use of the lozenge over a one-week period.

DETAILED DESCRIPTION:
This randomized, placebo controlled, double-blind, crossover study will use gas chromatography (GC) and oral microbial measurements to evaluate the reduction and control of intra-oral halitosis by an investigational lozenge containing the enzyme polyphenol oxidase and green coffee extract compared to a placebo control lozenge. A one-week washout period will precede the first crossover period and a one-week washout period will be implemented between periods 1 and 2. The study will consist of five study visits: Screening Visit, Period 1 Baseline Visit, Crossover Period 1 Day 8 Visit, Period 2 Baseline Visit, Crossover Period 2 Day 8 Visit.

ELIGIBILITY:
To be eligible for study participation, subjects must meet the following criteria:

Inclusion criteria:

1. Generally healthy males and females ≥18 years of age.
2. Able to read, sign and receive a copy of the signed informed consent form.
3. Have an average OralChroma™ reading ≥ 125 ppb hydrogen sulfide (H2S gas), volatile sulfur compound (VSC), based on 2 VSC measurements at Screening (Visit 1) and Baseline (Visit each 2 and 4), at least 12 hours after eating or drinking or oral hygiene.
4. Difference of the hydrogen sulfide gas readings is ≤ 500 ppb following the two mouth air samples for each VSC measurement for Screening (Visit 1) and Baseline (Visits 2 and 4).
5. Intra-oral cause of bad breath (non-systemic origin) as determined by health history or exam.
6. Have at least 18 natural teeth.
7. Agree to abstain from eating, drinking, breath mints, chewing gum, and any oral hygiene for at least 12 hours prior to evaluation of oral malodor at Screening, Baseline and Day 8 visits.
8. Agree to avoid drinking alcohol beverages and eating spicy foods, garlic and onions, cabbage, spices, cauliflower, and radishes (sulfur compounds) 48 hours prior to each study visit.
9. Agree to refrain from tongue brushing/cleaning for the duration of the study.
10. Adequate oral hygiene and no signs of oral neglect.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. History of allergy or significant adverse effects following use of oral hygiene products such as toothpastes, mouth rinses, breath mints, lozenges, or chewing gum or their ingredients.
2. History of allergies to ingredients in the test product.
3. Self-reported as pregnant or nursing.
4. Self-reported serious medical conditions.
5. Based on history and clinical exam: advanced and/or untreated periodontitis, frank caries, and mucosal diseases.
6. Antibiotic or anti-inflammatory medication within 30 days of screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Immediate Total Volatile Sulphur Compounds (T-VSC) | The change in T-VSCs from baseline to 5-minutes post-product assessment
  The primary efficacy endpoint is the immediate (no later than 5 minutes after dissolution of the lozenge) T-VSCs at Day 1 based on OralChroma™ measurement.

SECONDARY OUTCOMES:
T-VSCs over time | The change in T-VSCs over time from baseline to 1 hour, 2 hours, 4 hours (Day 1), and 7 days post-product assessments
  T-VSCs over time, based on OralChroma™ following daily product use
Specific VSCs over time | The change in specific VSCs over time from baseline to 1 hour, 2 hours, 4 hours (Day 1), and 7 days post-product assessments
  VSCs components [Hydrogen Sulfide (H2S), Methyl Mercaptan (CH3SH), and Dimethyl Sulfide (CH3SCH3) gases] over time following daily product use
Questionnaire | Day 1 and Day 8
  Post-product use questionnaire
Oral microbiome composition | Day 1 (pre and immediate post-product use, 5 minutes) and Day 8
  Microbiome profile by 16S rRNA sequencing, saliva and tongue biofilm samples collected

OTHER OUTCOMES:
Incidence of adverse events | Day 1 (4 hours) and Day 8
  Interviews to determine adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Holz, PhD, Study Director — Novozymes A/S
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No